CLINICAL TRIAL: NCT04240769
Title: Identifying the Trajectory of Normal Recovery Following Knee Arthroplasty Through Physical Activity Monitoring Via Wrist-Worn Accelerometry
Brief Title: Physical Activity Levels During Recovery Following Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 260855; 19/SW/0151 (Other: NHS Health Research Authority)
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: physical activity; rehabilitation; accelerometry
MeSH Terms: conditions — Motor Activity | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee Arthroplasty Patient: Patients undergoing primary total or unicompartmental knee arthroplasty for treatment of end-stage osteoarthritis.
  Interventions: Device: Total or Partial Knee Arthroplasty

INTERVENTIONS:
Device: Total or Partial Knee Arthroplasty — Reconstruction of part or all of the native articulation at the knee joint via implant.
  Other Names: Knee Replacement

SUMMARY:
The goal of this study is to utilize physical activity monitoring to determine the trajectory of normal recovery as it relates to a patient's ability to get up and get moving. From this work, we hope to be able to define the range in patients' physical activity following knee replacement surgery, and thus, give clinicians a tool and the methodology to identify patients whose recovery is not progressing as quickly as expected. Data from physical activity monitors will allow the research team to identify how active patients are, how vigorous that activity is, and how well that activity correlates with standard and commonly used patient questionnaires.

DETAILED DESCRIPTION:
This study is an observational study of the physical activity levels of adults who have been diagnosed with end-stage osteoarthritis of the knee and are undergoing knee replacement surgery at the Nuffield Orthopaedic Centre, Oxford. Data regarding patient activity and functional recovery will be collected using two methods. First, data will be collected through the extraction of three-axis accelerometer data, collected via a wrist-worn (and hip-worn for a subset of patients) physical activity monitor. This data will be collected in three intervals: pre-operatively, immediately postoperatively, and at 6 months postoperatively. Secondly, data will be collected by standard clinical assessment and patient reported outcome measures. These assessments will again take place pre-operatively, at 6 weeks postoperatively, and at 6 months postoperatively. Additional data will be collected through a simple activity diary, which asks the participants to log their monitor wear-time along with the times that they took bicycle rides or extended walks.

The expected duration of patient involvement is up to a total of 8 to 8.5 weeks over the course of up to 7 months. There are no clinical visits within this protocol beyond what is already within normal patient care. Patients will be asked to post their monitor back to the research centre for data collection and data processing twice during the study period.

The aim of this study is to assess the trajectory of recovery in terms of physical activity in the post-operative knee replacement population, and subsequently to define the expected path of early recovery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with required late stage osteoarthritis, undergoing knee arthroplasty in the next 3 months.
* In Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who are enrolled in another research study involving an investigational product or methodology that could alter physical activity.
* Participants are undergoing a revision arthroplasty surgery on the operative knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients undergoing primary total or unicompartmental knee arthroplasty for treatment of end-stage osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity | Physical activity will be evaluated for 7 days at approximately 2 weeks before surgery, for 6 continuous weeks immediately postoperatively and (for a subset of participants) for 7 continuous days at 6 months postoperatively.
  The primary outcome measure will physical activity, as extracted from analysis of raw accelerometer data from the activity monitor. Several variables will be extracted from the raw data, including average acceleration vector (Euclidean norm minus one), bouts of physical activity and percentage of active and sedentary time.

SECONDARY OUTCOMES:
Change in Oxford Knee Score | Pre-operative (baseline), 6 weeks, 6 months
  A patient reported outcome measure to assess patient benefit [Range 0 to 48, higher scores corresponding to better outcomes].
Change in EQ-5D-5L | Pre-operative (baseline), 6 weeks, 6 months
  A patient reported outcome measure to assess patient benefit. As summary index score from 0 to 1 is given, where 0 is the health state equivalent to dead, 1 is a full healthy outcome, and negative indicates a health state worse than dead. The score is derived from five sections (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression) scored 1 to 5, with higher corresponding to better outcomes. A second visual analogue score for perceived health is reported from 0 to 100 with higher scores indicating better perceived overall health.
Change in University of California, Los Angeles (UCLA) Activity Score | Pre-operative (baseline), 6 weeks, 6 months
  A self-reported score to assess patient benefit and physical activity. The score ranges from 1 to 10 where higher scores indicate greater levels of physical activity
Change in International Physical Activity Questionnaire Questionnaire - Short Form | Pre-operative (baseline), 6 weeks, 6 months
  A self-reported score to assess patient benefit and physical activity. The score can be reported in one of three categories: Low, Moderate, or High physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Small, MS, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford University Hospitals Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available within 6 months following study completion.
Access Criteria: Data access requests will be reviewed by the trial steering committee.